CLINICAL TRIAL: NCT06712784
Title: Supporting Patients With Autism Spectrum Disorder (ASD) During Needle-related Hospital Visits Through the Use of Behavior Analytic Strategies
Brief Title: Behavior Analytic Support of Needle-related Hospital Visits for Autistic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-45181
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Behavior analytic research; Needle-related healthcare visits; Simulation visits; Differential reinforcement of alternative behavior (DRA)
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Packet (Experimental): 3-5 autistic BMC patients who have a history of engaging in challenging behaviors during needle-related procedures who are able to attend simulation sessions at BMC at least 2 times per month. A caregiver and clinician will also be recruited for each child participant.
  Interventions: Behavioral: Treatment Package (for both simulation and procedure sessions

INTERVENTIONS:
Behavioral: Treatment Package (for both simulation and procedure sessions — Treatment Package for both simulation and procedure sessions will include visit priming (contingency specifying stimuli in the form of social stories and YouTube videos) and differential reinforcement of alternative behavior (DRA).

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the behavior analytic intervention in reducing the number of challenging behaviors exhibited by patients with Autism Spectrum Disorder (ASD) while increasing compliance with needle-related simulations and procedures. A second purpose is to assess the social validity of this study as evidenced by patient and/or caregiver acceptability. The study wil take place at Boston Medical Center (BMC).

A Single Subject Design (SSD) wil be utilized as it allows for detailed, individualized assessment of how interventions affect behavior over time in this type of behavior analytic research. By focusing on each participant as an individual and having each participant act as their own control, it demonstrates clear cause-and-effect relationships, showing how behavior changes with the introduction or withdrawal of an intervention. This method is flexible, enabling ongoing adjustments to treatments based on real-time data, making it particularly useful in personalized interventions and ensuring effectiveness for patients with unique needs such as those who would be eligible to enroll and participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of autistic patients who have been historically engaged in challenging behaviors during needle-related procedures at a Boston Medical Center (BMC)
* Established BMC autistic patients (ages 3+) who have a history of engaging in challenging behaviors in the presence of needle-related medical stimuli.
* BMC Medical Providers (i.e., phlebotomists, medical doctors, registered nurses, certified nursing assistants, registered dieticians, and medical assistants) who either: 1) order needle-related medical procedures for participants to be conducted during procedure visits and/or 2) are present to conduct the ordered procedure
* English speaking participants

Exclusion Criteria:

* Patients who are unable to visit BMC a minimum of 2 times per month
* No history of challenging behaviors in medical appointments involving the presentation of needle(s)
* Patients and caregivers who do not speak English or are unable to utilize interpreter services to complete assessments and surveys

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have a decrease in challenging behaviors in the presence of medical stimuli (needles) | Baseline, on average 4 months
  A challenging behavior is defined as one that is either harmful, disruptive, or difficult to manage as documented on an investigator-developed task list.
Number of task list steps completed in the absence of challenging behaviors | Baseline, on average 4 months
  This will be assessed using the investigator-developed task list.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline McKendry, MS BCBA LABA, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No